CLINICAL TRIAL: NCT04508426
Title: A Phase 1, Absorption, Metabolism, and Excretion Study of [14C]AR882 Orally Administered to Healthy Adult Male Subjects
Brief Title: Single-dose AME Study With [14C]AR882 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR882-103
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mass Balance (Experimental)
  Interventions: Drug: [14C]AR882

INTERVENTIONS:
Drug: [14C]AR882 — Single dose of [14C]AR882

SUMMARY:
This is an open-label, single-dose, absorption, metabolism, excretion, and mass balance study following a single dose of [14C]AR882 in healthy adult male subjects. Whole blood, plasma, urine, and fecal samples will be analyzed for at least 144 hours following the single dose of AR882 to measure total radioactivity and plasma drug concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Body weight no less than 50 kg and body mass index (BMI) within the range of ≥ 18 and ≤ 33 kg/m2
* Must have a minimum of 1 bowel movement every 2 days
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs

Exclusion Criteria:

* Inadequate venous access or unsuitable veins for repeated venipuncture
* Positive serology to HIV (HIV1 and HIV2) and/or Hepatitis C antibodies, and/or Hepatitis B

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Total radioactivity (TRA) in urine | Days 1-14
TRA in feces | Days 1-14
TRA concentration equivalents in plasma | Days 1-14
TRA concentration equivalents in whole blood | Days 1-14
Area under the curve (AUC) for plasma [14C]-AR882 | 7 Days
  Profile from plasma in terms of AUC following a single dose of [14C]-AR882
Time to maximum plasma concentration (Tmax) for [14C]-AR882 | 7 Days
  Profile from plasma in terms of Tmax following a single dose of [14C]-AR882
Maximum plasma concentration (Cmax) for [14C]-AR882 | 7 Days
  Profile from plasma in terms of Cmax following a single dose of [14C]-AR882
Apparent terminal half-life (t1/2) for [14C]-AR882 | 7 Days
  Profile from plasma in terms of t1/2 following a single dose of [14C]-AR882

SECONDARY OUTCOMES:
Incidence of Adverse Events, changes in laboratory, electrocardiogram, and vital signs [14C]-AR882 | Days 1-14

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No